CLINICAL TRIAL: NCT04984980
Title: Efficacy and Safety of the Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab in Initially Unresectable Biliary Tract Cancer
Brief Title: Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab in Unresectable Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-176-2096
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Biliary Tract Carcinoma; Initially Unresectable
MeSH Terms: interventions — Oxaliplatin; sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab Gemcitabine: 1000mg/m^2, iv, d1, d8, q3w Oxaliplatin: 100mg/m^2, iv, d1, q3w Sintilimab: 200mg, iv, d1, q3w Bevacizumab: 5mg/kg, d1, q3w
  Interventions: Drug: Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab

INTERVENTIONS:
Drug: Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab — Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab

SUMMARY:
Study design: Prospective, single-arm, single-center phase II clinical study; Primary endpoint: Conversion rate; Secondary endpoints: Safety, disease control rate, disease-free survival, and overall survival; Main characteristics of enrolled patients: Patients with initially unresectable biliary tract cancer; Interventions: Combination of Gemcitabine, Oxaliplatin, Sintilimab and Bevacizumab; Sample size: 34 patients; Treatment until: 1. successfully conversed to resectable disease 2. progressed disease 3. intolerable toxicity 4. patient requests withdrawal; Research process: In this study, patients who met the inclusion criteria were evaluated at the end of every 3 weeks of treatment, up to surgical treatment or disease progression; Safety evaluation: Evaluate adverse reactions according to CTCAE 4.0; Follow up: 12 months after the last case was enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years;
2. ECOG 0~1;
3. Histologically or cytologically confirmed carcinoma of the bile duct or gallbladder;
4. Imaging assessment of disease stage III/IVA/any TN1M0*;
5. The main organs have good functions and the examination indexes meet the following requirements:
6. Blood routine test:

   Hemoglobin ≥90 g/L (no blood transfusion within 14 days); Neutrophils count ≥1.5×10^9/L; Platelet count ≥80×10^9/L;
7. Biochemical tests:

   Total bilirubin ≤2×ULN (upper limit of normal value); Blood alanine aminotransferase (ALT) or blood aspartate aminotransferase (AST) ≤ 2.5×ULN; Endogenous creatinine clearance rate ≥ 50 mL /min (Cockcroft-Gault formula);
8. Voluntarily signed the informed consent;
9. Good compliance and family members are willing to cooperate with follow-up.

Exclusion Criteria:

1. Other uncured malignancies;
2. Pregnant or lactating women, if the subject becomes pregnant during the study period, should withdraw from the clinical trial;
3. Previous anti-tumor therapy for the disease in this study;
4. Participated in other drug clinical trials within one month;
5. Patients with known history of other systemic serious diseases before screening;
6. Long-term unhealed wounds or incomplete healed fractures;
7. Have a history of organ transplantation;
8. Abnormal blood coagulation, with bleeding tendency (14 days before randomization must meet: INR within the normal range without the use of anticoagulants); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogs; The use of low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (not more than 100 mg daily) for prophylactic purposes is permitted, provided that INR is less than 1.5;
9. The incidence of arterial/venous thrombosis events in the previous year, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism, was screened;
10. People with a history of psychotropic substance abuse and unable to get rid of it or with mental disorders; Have a history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;

12. Concomitant diseases that, in the Investigator's judgment, seriously endanger patient safety or affect patient completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 3 weeks
  objective response rate

SECONDARY OUTCOMES:
Safety：the incidence of adverse events and serious adverse events | 3 weeks
  Incidence of adverse events and serious adverse events
disease control rate | 3 weeks
  disease control rate
progress-free survival | 3 weeks
  progress-free survival
overall survival | 3 weeks
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China